CLINICAL TRIAL: NCT06521905
Title: Prospective, Multicenter, Randomized Controlled Study on the Treatment of Stent Underexpansion Caused by Calcification Using Intravascular Lithotripsy
Brief Title: Clinical Trial on the Treatment of Stent Underexpansion Caused by Calcification Using Intravascular Lithotripsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Kefei Dou, MD, Professor, China National Center for Cardiovascular Diseases, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: intravascular lithotripsy
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Intravascular Lithotripsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): intravascular lithotripsy is used on the basis of high-pressure balloon dilation
  Interventions: Device: intravascular lithotripsy
- control group (Active Comparator): only use more positive high-pressure ballon dilation
  Interventions: Device: high-pressure ballon

INTERVENTIONS:
Device: intravascular lithotripsy — The intravascular lithotripsy can intermittently release acoustic pressure waves at the site of vascular calcification lesions, thereby achieving the goal of rupturing calcified plaques; After the rupture of calcified plaques, the vascular calcification lesions can be fully dilated with the help of lower balloon inflation pressure.
  Arms: experimental group
Device: high-pressure ballon — High pressure balloon dilation, as the main method for traditional treatment of insufficient stent expansion caused by calcification, has a good therapeutic effect on insufficient stent expansion caused by calcification
  Arms: control group

SUMMARY:
Our aim is to investigate the efficacy and safety of intravascular lithotripsy(IVL) in the treatment of stent underexpansion caused by calcification through a prospective, multicenter, randomized controlled trial. Patients with inadequate stent expansion due to calcification detected by intravascular ultrasound(IVUS) were randomly divided into two groups. The experimental group received IVL in addition to high-pressure balloon post-dilation, while the control group only received high-pressure balloon post-dilation. Follow up for 1 year is conducted to determine the safety and efficacy of IVL application based on the primary efficacy endpoint, key secondary efficacy endpoint, other secondary efficacy endpoint, and safety endpoint.

DETAILED DESCRIPTION:
In order to investigate the effectiveness and safety of intravascular lithotripsy(IVL) in patients with calcium induced stent insufficiency, we designed a prospective, randomized, controlled, single blind, multicenter, and superior efficacy clinical trial. We include a real-world population of patients who had stent underexpansion due to calcification detected by intravascular ultrasound(IVUS) in the target vessel after percutaneous coronary intervention(PCI) and met the inclusion and exclusion criteria. In addition to routine clinical treatment, IVUS testing was performed on patients after PCI. Patients who met the criteria for stent underexpansion detected by IVUS are randomly divided into two groups. The experimental group received IVL intervention on the basis of high-pressure balloon post-dilation, while the control group received more aggressive high-pressure balloon post-dilation treatment. The satisfaction rate of stent dilation detected by IVUS in both groups after IVL or high-pressure balloon post-dilation was taken as the main efficacy endpoint. MACE events (composed of cardiovascular death, target vessel myocardial infarction and target vascular revascularization) from PCI to one-year follow-up are evaluated. And the acquisition of lumen after treatment is used as other secondary efficacy endpoints. We use postoperative complications such as coronary artery spasm, dissection, acute occlusion, and persistent ventricular arrhythmia as safety endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-80 years old, male or non pregnant female
2. The patient or guardian can voluntarily sign and understand the informed consent form, and can accept follow-up
3. Asymptomatic ischemic, stable or unstable angina or myocardial infarction (MI) (including ST segment elevation and non ST segment elevation MI) with chest pain onset to hospital admission time>24 hours, as well as old myocardial infarction patients
4. Visually assess the target lesion with a reference vessel diameter of 2.5-4.0mm, diameter stenosis degree ≥ 70% or ≥ 50%, and evidence of ischemia
5. The target lesion is the only lesion that requires treatment this time
6. Patients suitable for percutaneous coronary stent implantation
7. Confirmed by coronary angiography or IVUS testing that the target lesion is calcified, with any degree of calcification
8. After surgical treatment for calcified lesions, IVUS testing confirmed that it meets the criteria for incomplete stent expansion

Exclusion Criteria:

Exclusion criteria for patient level:

1. Individuals with abnormal coagulation function tests
2. Patients with severe hemodynamic disorders
3. Clinical manifestations of heart failure with LVEF<30%
4. I have experienced an acute myocardial infarction in the past week
5. Patients allergic to heparin, contrast agents, antiplatelet drugs, anticoagulants, anesthetics, etc
6. Patients with severe myocardial bridge/negative remodeling or target vessel thrombosis
7. Pregnant or lactating women
8. Patients with malignant tumors or comorbidities with a life expectancy of less than 12 months
9. History of active peptic ulcer or gastrointestinal bleeding within 6 months prior to enrollment
10. Stroke occurred within 6 months prior to enrollment, excluding transient ischemic attack (TIA) and cerebral infarction
11. Severe liver and kidney function impairment, transaminase levels exceeding the upper limit of normal by more than three times, creatinine levels greater than 2.5mg/dL (221 μ moI/L), or chronic renal failure requiring long-term dialysis
12. Anti thrombotic therapy intolerance
13. Severe anemia, thrombocytopenia, or leukopenia
14. History of severe bleeding (intracranial, gastrointestinal)
15. Also participating in other patients who have not completed clinical trials at the same time
16. Patients with poor compliance and inability to complete the study on time
17. Other situations deemed unsuitable by researchers to participate in this clinical study

Exclusion criteria for vascular level:

1. Thrombotic lesion
2. Bridge vascular disease
3. Angiography shows tortuous vascular pathways, making it difficult for experimental instruments to reach the target position or retrieve them

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction Rate of Stent Expansion[Effcacy] | immediately after percutaneous coronary intervention(PCI)
  Satisfied stent expansion is defined as meeting the standard of good expansion after stent implantation through IVUS after PCI

SECONDARY OUTCOMES:
Major Cardiovascular Events[Effcacy] | 1 year after after percutaneous coronary intervention(PCI)
  a composite endpoint of cardiovascular death, target vessel myocardial infarction and target vessel revascularization
Lumen Obtainment after PCI[Effcacy] | immediately after percutaneous coronary intervention(PCI)
  changes in lumen area after treatment
Incidence of Treatment-Emergent Complications[Safety] | immediately after percutaneous coronary intervention(PCI)
  Postoperative complications such as coronary spasm, dissection, acute occlusion, persistent ventricular arrhythmia, etc

CONTACTS AND LOCATIONS:
Overall Officials: Kefei Dou, Doctor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital

IPD SHARING:
Plan to Share IPD: No
Except for privacy data, all other data can be made public